CLINICAL TRIAL: NCT01625689
Title: Assessment of the Safety and Immunogenicity of a Single Dose of Intranasal Seasonal Trivalent Live-Attenuated Influenza Vaccine Among Children Aged 24 Through 59 Months in Bangladesh
Brief Title: Safety and Immunogenicity of a Single Dose of Intranasal Seasonal Trivalent Live-Attenuated Influenza Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PATH Vaccine Solutions (Other)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Organization: PATH (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LAIV-BD-01
Record Dates: First submitted 2012-06-14; First posted 2012-06-21 (Estimated); Results first posted 2015-06-01 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2012-06

CONDITIONS: Influenza
Keywords: Influenza vaccines; Influenza, Human; Live Attenuated Influenza Vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SIIL LAIV (Experimental): SII LAIV is a live, trivalent seasonal influenza vaccine. The viral strains in seasonal trivalent influenza vaccine (human, live attenuated) are antigenically similar to A/California/7/2009 (H1N1), A/Perth/16/2009 (H3N2) and B/Brisbane/60/2008 Type B, as per the WHO recommended strains for the Northern hemisphere 2011-12 influenza season
  Interventions: Biological: SIIL LAIV (live, trivalent seasonal influenza vaccine)
- Placebo (Placebo Comparator): Placebo identical in appearance to experimental vaccine.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: SIIL LAIV (live, trivalent seasonal influenza vaccine) — Dose: 0.5 mL, The viral strains in seasonal trivalent influenza vaccine (human, live attenuated) are antigenically similar to A/California/7/2009 (H1N1), A/Perth/16/2009 (H3N2) and B/Brisbane/60/2008 Type B, as per the WHO recommended strains for the Northern hemisphere 2011-12 influenza season
  Arms: SIIL LAIV
Biological: Placebo — Inactive placebo will be identical to SII LAIV in appearance, ingredients, and concentrations, except it will be missing attenuated influenza virus.
  Arms: Placebo

SUMMARY:
In this Phase II randomized controlled clinical trial, generally healthy male and female children from 24 through 59 months of age will be enrolled in Kamalapur (Dhaka), Bangladesh. The study is expected to continue for at least 6 months following vaccination. The experimental intervention is Serum Institute of India Ltd's Trivalent, Seasonal Live Attenuated Influenza Vaccine (SIIL LAIV). The study vaccine has been formulated according to WHO recommendations for the 2011-2012 Northern Hemisphere influenza season. The SIIL LAIV is administered in a 0.5 ml intranasal dose (one spray of 0.25 ml per nostril) via a reusable sprayer device and a single-use nozzle that produces a fine mist that is primarily deposited in the nose and nasopharynx. The comparator vaccine will be an inactive placebo identical in appearance to the active vaccine.

The primary study hypothesis is that LAIV is safe and well tolerated by children aged 24 through 59 months in Bangladesh. A secondary hypothesis is that LAIV is immunogenic among children receiving study vaccine as compared to children receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female child at least 24 months of age and no older than 59 months of age at the time of study vaccination
* A child whose parent or guardian's primary residence, at the time of study vaccinations, is within the Kamalapur surveillance site catchment area and who intends to be present in the area for the duration of the trial
* A child whose parent or legal guardian is willing to provide written informed consent prior to the participant's study vaccination

Exclusion Criteria:

* Has any serious chronic disease including progressive neurologic disease, tuberculosis, Down's syndrome or other cytogenetic disorder, or known or suspected disease of the immune system
* Is receiving immunosuppressive agents including systemic corticosteroids during the two weeks prior to study vaccination
* Has a history of documented hypersensitivity to eggs or other components of the vaccine (including gelatin, sorbitol, lactalbumin and chicken protein), or with life-threatening reactions to previous influenza vaccinations
* Is receiving aspirin therapy or aspirin-containing therapy currently or two weeks before
* Lives in household with somebody currently participating in a respiratory vaccination or antiviral study
* Has current or past participation (within 2 months of trial enrollment visit) in any clinical trial involving a drug or biologic with activity against respiratory disease
* Has any condition determined by investigator as likely to interfere with evaluation of the vaccine or be a significant potential health risk to the child

Ages: 24 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 309 (Actual)
Dates: Start 2012-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W. Abdullah Brooks, MD, MPH, Principal Investigator — JHSPH, ICDDR,B
Locations (1):
- ICDDR,B Kamalapur, Dhaka, Bangladesh

REFERENCES:
- [Derived] Lewis KDC, Ortiz JR, Rahman MZ, Levine MZ, Rudenko L, Wright PF, Katz JM, Dally L, Rahman M, Isakova-Sivak I, Ilyushina NA, Matyushenko V, Fry AM, Lindstrom SE, Bresee JS, Brooks WA, Neuzil KM. Immunogenicity and Viral Shedding of Russian-Backbone, Seasonal, Trivalent, Live, Attenuated Influenza Vaccine in a Phase II, Randomized, Placebo-Controlled Trial Among Preschool-Aged Children in Urban Bangladesh. Clin Infect Dis. 2019 Aug 16;69(5):777-785. doi: 10.1093/cid/ciy1003. PMID 30481272
- [Derived] Brickley EB, Wright PF, Khalenkov A, Neuzil KM, Ortiz JR, Rudenko L, Levine MZ, Katz JM, Brooks WA. The Effect of Preexisting Immunity on Virus Detection and Immune Responses in a Phase II, Randomized Trial of a Russian-Backbone, Live, Attenuated Influenza Vaccine in Bangladeshi Children. Clin Infect Dis. 2019 Aug 16;69(5):786-794. doi: 10.1093/cid/ciy1004. PMID 30481269

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 309 participants were consented and enrolled in the study. 9 participants were ineligible to receive study vaccination. 300 total participants were vaccinated and followed through the study period.
Groups:
- Serum Institute of India, Ltd. (SIIL) LAIV: The Serum Institute of India, Ltd. (SIIL) live attenuated influenza vaccine (LAIV) (human, live attenuated, trivalent seasonal influenza vaccine): The viral strains in are antigenically similar to A/California/7/2009 (H1N1), A/Perth/16/2009 (H3N2) and B/Brisbane/60/2008 Type B, as per the WHO recommended strains for the Northern hemisphere 2011-12 influenza season
- Placebo: Inactive placebo was identical to SIIL LAIV in appearance, ingredients, and concentrations, except it was missing attenuated influenza virus.
Period: Overall Study
Arm/Group | Serum Institute of India, Ltd. (SIIL) LAIV | Placebo
Started | 150 | 150
Completed | 148 | 149
Not Completed | 2 | 1
Not completed — Migration | 2 | 1

BASELINE CHARACTERISTICS:
Population: All participants enrolled who received a single dose of LAIV or placebo.
Groups:
- SIIL LAIV: The SIIL LAIV (human, live attenuated, trivalent seasonal influenza vaccine): The viral strains in are antigenically similar to A/California/7/2009 (H1N1), A/Perth/16/2009 (H3N2) and B/Brisbane/60/2008 Type B, as per the WHO recommended strains for the Northern hemisphere 2011-12 influenza season
- Placebo: Inactive placebo was identical to the SIIL LAIV in appearance, ingredients, and concentrations, except it was missing attenuated influenza virus.
- Total: Total of all reporting groups
Arm/Group | SIIL LAIV | Placebo | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 150 | 150 | 300
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 66 | 139
  Male | 77 | 84 | 161
Region of Enrollment [Number; unit: participants]
  Bangladesh | 150 | 150 | 300

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs), All-cause Hospitalizations, and Protocol-defined Wheezing Illness (PDWI) Episodes
Description: PDWI: Participants meeting illness criteria, seeking care in health facility, and with wheeze identified by a study physician
  Illness criteria: The presence of one Category A (Fever (>=38°C), tachypnea, danger signs (chest-indrawing, lethargy, cyanosis, inability to drink, convulsions), difficult breathing, noisy breathing, ear pain or discharge) or two Category B findings (Cough, rhinorrhea, sore throat, myalgia/arthralgia, chills, headache, irritability/decreased activity, vomiting)
  Wheeze: Long high-pitched whistling or musical sound on expiration heard by auscultation
Time Frame: 6 months following vaccination
Population: Safety analysis population
Measure: Number; unit: participants
Groups:
- Placebo: Inactive placebo was identical to SII LAIV in appearance, ingredients, and concentrations, except it was missing attenuated influenza virus.
Arm/Group | SIIL LAIV | Placebo
Number analyzed (Participants) | 150 | 150
participants
  Serious Adverse Events | 6 | 0
  Protocol Defined Wheezing Illness (PDWI) | 13 | 16
  Hospitalizations | 3 | 0

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs), All-cause Hospitalizations, and Protocol-defined Wheezing Illness (PDWI) Episodes
Description: as for outcome 1
Time Frame: 42 days following vaccination
Reporting Status: Not Posted

3. Primary Outcome: Percentage of Participants With Unsolicited Adverse Events (AEs)
Time Frame: Throughout study period, through at least 6 months following vaccination
Measure: Number; unit: percentage of participants
Arm/Group | SIIL LAIV | Placebo
Number analyzed (Participants) | 150 | 150
percentage of participants
  Diarrheal Illness | 25.3 | 21.3
  Oral thrush | 17.3 | 12.0
  Boil/abscess/skin infection/ulcer/cyst | 7.3 | 12.0
  Helminthiasis | 6.0 | 7.3
  Scabies | 5.3 | 4.0
  Abdominal pain/distension | 3.3 | 4.0
  Allergy | 4.0 | 4.0
  Fungal Infection | 4.0 | 3.3
  Other | 36.7 | 34.0

4. Primary Outcome: Percentage of Participants With Solicited Local and Systemic Reactions
Description: Local reactions: Nasal discomfort, Runny nose, Stuffy nose, Sneezing, Ear pain
  Systemic Reactions: Cough, Headache, Loss of Appetite, Fever, Irritability, Nausea, Sore throat, Lethargy
Time Frame: Through 7 days following vaccination
Population: Safety analysis population
Measure: Number; unit: percentage of participants
Arm/Group | SIIL LAIV | Placebo
Number analyzed (Participants) | 150 | 150
percentage of participants
  Measured fever (>=38.0) | 3.3 | 3.3
  Ear pain | 1.3 | 1.3
  Cough | 6.7 | 5.3
  Runny nose/nasal congestion | 20.7 | 22.7
  Sore throat | 1.3 | 0.0
  Headache | 0.7 | 0.0
  Irritability/decreased activitity | 0.0 | 0.0
  Vomiting | 1.3 | 2.0
  Lethargy | 0.0 | 0.0
Statistical Analysis 1: Comparison: SIIL LAIV vs Placebo; Test type: Superiority or Other; p >= 0.498, Fisher Exact — No comparison between the LAIV and placebo groups by type of solicited reaction had a p-value below 0.498

5. Secondary Outcome: The Post-vaccination Anti-influenza Immunologic Response Will be Measured Based on the Type of Immunologic Assay and Categorized by Vaccine Virus Strain, Participant Baseline Serostatus, and Vaccine Allocation
Time Frame: Approximately 21 days post-vaccination
Reporting Status: Not Posted

6. Secondary Outcome: Post Vaccination SIIL LAIV Virus Shedding/Vaccine-take Will be Parameterized by the Percentage of Participants With Detectable Virus by Post Vaccination Day.
Time Frame: 2, 4, and 7 days post-vaccination
Reporting Status: Not Posted

7. Secondary Outcome: Clinical Characteristics of Influenza, Including Influenza Coinfections With Other Bacterial and Viral Respiratory Pathogens, Will be Parameterized as the Percentage of Participants Categorized by Vaccine Allocation
Time Frame: 6 months post-vaccination
Reporting Status: Not Posted

8. Secondary Outcome: Viral Etiologies of Acute Respiratory and Febrile Illness Will be Parameterized as the Percentage of Those With Each Particular Laboratory-confirmed Respiratory Virus Infection Categorized by Vaccine Allocation
Time Frame: 6 months post-vaccination
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Throughout study period, through at least 6 months post-vaccination.
Arm/Group | SIIL LAIV | Placebo
Serious Adverse Events (participants affected / at risk) | 6/150 | 0/150
Other Adverse Events (participants affected / at risk) | 96/150 | 94/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SIIL LAIV (N=150) | Placebo (N=150)
Traumatic Injury/fracture/overdose (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
abdominal pain/gastroenteritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SIIL LAIV (N=150) | Placebo (N=150)
diarrheal illness (Gastrointestinal disorders) | 38 | 32
Oral thrush (Infections and infestations) | 26 | 18
Boil/Abscess/skin infection/ulcer/cyst (Infections and infestations) | 11 | 18
Helminthiasis (Infections and infestations) | 9 | 7
Scabies (Infections and infestations) | 8 | 6
Abdominal pain/distension (Gastrointestinal disorders) | 5 | 6
Allergy (General disorders) | 6 | 6
Fungal Infection (Infections and infestations) | 6 | 5
Other (Infections and infestations) | 55 | 51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less